CLINICAL TRIAL: NCT05673200
Title: Phase I Study Targeting DNA Methyltransferases in Metastatic Triple-Negative Breast Cancer
Brief Title: Testing the Addition of an Anti-cancer Drug, ASTX727 (Cedazuridine, Decitabine), to Chemotherapy (Paclitaxel) and Immunotherapy (Pembrolizumab) for Metastatic Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-10810; NCI-2022-10810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10546 (Other: Dana-Farber - Harvard Cancer Center LAO); 10546 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Unresectable Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; Specimen Handling; decitabine and cedazuridine drug combination; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ASTX727, paclitaxel, pembrolizumab) (Experimental): Patients receive ASTX727 PO on days 1-5, 1-4, 1-3, or days 1, 3, and 5 of each cycle, and paclitaxel IV over 1 hour on days 1, 8, and 15 of each 28-day cycle or days 1 and 8 of each 21-day cycle. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV over 30 minutes every 6 weeks (treatment day varies in 28-day cycles; day 1 of every odd 21-day cycle) in the absence of disease progression or unacceptable toxicity. Patients undergo collection of blood samples and CT and/or MRI throughout the trial. Patients in the dose-expansion phase also undergo a tumor biopsy during screening and day 1 of the treatment cycle 2 of the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Decitabine and Cedazuridine; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Biological: Pembrolizumab

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of ASTX727 when given in combination with a usual approach of treatment with paclitaxel and pembrolizumab in patients with triple-negative breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic). The usual approach is defined as care most people get for this type of cancer. The usual approach for patients with metastatic triple negative breast cancer who are not in a study is chemotherapy with drugs like paclitaxel, carboplatin, cisplatin, eribulin, vinorelbine, capecitabine, gemcitabine, doxorubicin or cyclophosphamide. There is a protein called PD-L1 that helps regulate the body's immune system. For patients who have PD-L1+ tumors, immunotherapy (pembrolizumab) is usually added to paclitaxel or carboplatin/gemcitabine as initial treatment. For patients who have PD-L1-negative tumors, chemotherapy alone is used, without immunotherapy. ASTX727 is a combination of two drugs, decitabine and cedazuridine. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Paclitaxel is in a class of medications called antimicrotubule agents. It stops tumor cells from growing and dividing and may kill them. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving ASTX727 with usual treatment approach with paclitaxel and pembrolizumab may be able to shrink or stabilize the tumor for longer than the usual approach alone in patients with metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of oral decitabine and cedazuridine (ASTX727) administered concurrently with paclitaxel and pembrolizumab (MK-3475). (Part 1 [Dose finding cohort]) II. To further describe the adverse event profile of the combination of oral ASTX727 at the RP2D when administered concurrently with paclitaxel and pembrolizumab (MK-3475). (Part 2 [Expansion cohort])

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity of this combination. II. To describe the adverse event profile of the combination of oral ASTX727 administered concurrently with paclitaxel and pembrolizumab (MK-3475). (Part 1 [Dose finding cohort]) III. To explore the association of baseline gene expression profiles (ribonucleic acid-sequencing [RNA-Seq]), with focus on DNMT isoforms and TRAF-6 signaling, with clinical benefit from study treatment, as well as changes in expression after 1 cycle of treatment. (Part 2 [Expansion cohort]) IV. To evaluate the impact of study treatment on methylation (in tumor tissue and circulating tumor deoxyribonucleic acid [ctDNA]). (Part 2 [Expansion Cohort])

EXPLORATORY OBJECTIVES:

I. To preliminarily evaluate the association of baseline DNMT3A protein expression by immunohistochemistry (IHC) and antitumor activity, as well as whether study treatment results in reduction of DNMT3A protein expression. (Part 1 [Dose finding cohort]) II. To preliminarily evaluate the association of baseline tumor-infiltrating lymphocytes (TILs) and PD-L1 expression with antitumor activity. (Part 1 [Dose finding cohort]) III. To evaluate the impact of study treatment on ctDNA methylation, peripheral blood immune phenotype and function, and serum thymidine kinase (TK1). (Part 1 [Dose finding cohort]) IV. To evaluate the impact of study treatment on immune phenotype (in tumor and peripheral blood) and function. (Part 2 [Expansion cohort]) V. To explore the impact of study treatment on immune-related genomic signaling by RNA-Seq. (Part 2 [Expansion cohort]) VI. To evaluate the association between baseline TILs and PD-L1 expression with treatment response, as well as changes in expression after 1 cycle of treatment. (Part 2 [Expansion cohort]) VII. To evaluate the association between mutations in driver genes, epigenetic genes and homologous recombination deficiency status (assessed by whole exome sequencing) with clinical outcome. (Part 2 [Expansion cohort])

OUTLINE: This is a dose-escalation study of ASTX727 in combination with fixed-dose pembrolizumab and fixed or reduced-dose paclitaxel, followed by a dose-expansion study.

Patients receive ASTX727 orally (PO) on days 1-5, 1-4, 1-3, or days 1, 3, and 5 of each cycle, and paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15 of each 28-day cycle or days 1 and 8 of each 21-day cycle. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV over 30 minutes every 6 weeks (treatment day varies in 28-day cycles; day 1 of every odd 21-day cycle) in the absence of disease progression or unacceptable toxicity. Patients undergo collection of blood samples and computed tomography (CT) and/or magnetic resonance imaging (MRI) throughout the trial. Patients in the dose-expansion phase also undergo a tumor biopsy during screening and day 1 of the treatment cycle 2 of the study.

Patients will be followed every 6 months for 3 years post registration or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed triple-negative breast cancer (TNBC) (estrogen receptor [ER] and progesterone receptor [PR] =< 10%, human epidermal growth factor receptor-2 [HER2]-negative per American Society of Clinical Oncology [ASCO]/College of American Pathologists [CAP] guidelines) that is metastatic or unresectable
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of ASTX727 in combination with pembrolizumab (MK-3475) and paclitaxel in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (or Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (within 14 days prior to registration)
* Platelets >= 100,000/mm^3 (within 14 days prior to registration)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (within 14 days prior to registration)

  * Criteria must be met without packed red blood cell (pRBC) transfusion within the prior 14 days of registration. Participants can be on stable dose of erythropoietin (90 days or more prior to registration)
* Creatinine clearance (CrCl) >= 30 mL/min (within 14 days prior to registration)

  * Glomerular filtration rate (GFR) can also be used in place of CrCl
* Total bilirubin =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 × ULN (within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 3 x institutional ULN (within 14 days prior to registration)
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if there is evidence of measurable extracranial disease, and if follow-up brain imaging 4 weeks after central nervous system (CNS)-direct therapy shows no evidence of progression. Patients with carcinomatous meningitis are not eligible.
* Patients with a prior malignancy whose natural history does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Concurrent use of other antineoplastic treatments is not allowed.
* Patients should be New York Heart Association Functional Classification of class II or better.
* Patients who have received live attenuated vaccines within the 30 days prior to registration are not eligible. Seasonal flu vaccines that do not contain live virus, and coronavirus disease 2019 (COVID-19) vaccinations and boosters are permitted.
* Patients with prior history of peripheral neuropathy are allowed if it has recovered to grade 1 or less.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial.
* Patients who have received 0-3 prior lines of chemotherapy in the metastatic setting. Patients who have received prior PD-1/PD-L1 monoclonal antibodies in any disease setting are eligible.
* For enrollment to Dose Finding Cohort: Availability and willingness to provide archival tumor tissue as required per protocol.
* For enrollment to Dose Expansion Cohort: (i) Willingness to provide baseline and 3-week tumor tissue biopsy specimens. (ii) Patients must have a measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* The effects of ASTX727 and pembrolizumab (MK-3475) on the developing human fetus are unknown. For this reason and because these agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 180 days after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Pregnant women are excluded from this study because pembrolizumab (MK-3475) is an anti PD-1 monoclonal antibody agent, ASTX727 is a hypomethylating agent, and paclitaxel is a class D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab (MK-3475), breastfeeding should be discontinued if the mother is treated with pembrolizumab (MK-3475). These potential risks may also apply to other agents used in this study. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 180 days after completion of study treatment.
* Ability to understand and the willingness to sign a written informed consent document (or have legally acceptable representative sign, if applicable).
* Patients who have recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia.

  * Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has not received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony-stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF], or recombinant erythropoietin) within 4 weeks prior to registration.

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within the 7 days prior to registration.
* Has a known additional malignancy that is progressing or requires active treatment.
* Has an active autoimmune disease that has required systemic treatment within 2 years prior to registration (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Current treatment with systemic steroids up to 10 mg of prednisone daily or equivalent is allowed.
* Patients with uncontrolled intercurrent illness (including but not limited to interstitial lung disease or active, non-infectious pneumonitis) or a history of (non-infectious) pneumonitis that required steroids.
* History of grade 3-4 immediate hypersensitivity reaction to paclitaxel or other drugs formulated in polyoxyl 35 castor oil.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ASTX727, pembrolizumab (MK-3475), and/or paclitaxel.
* Has a known history of active tuberculosis (TB).
* Gastrointestinal disorder that may impact absorption of oral medications.
* History of solid organ or bone marrow transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2027-02-23 (Estimated); Study Completion 2027-02-23 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) of ASTX727 in combination with paclitaxel and pembrolizumab (MK-3475) (Dose Finding Phase) | Within the first cycle of treatment (28 days)
  Defined as the highest dose level among those under consideration where at most 1 of 6 patients develops a dose limiting toxicity and 2 or more of the 3-6 patients treated at the next higher dose level develop a dose limiting toxicity.
Safety profile of ASTX727 in combination with paclitaxel and pembrolizumab (MK-3475) (Dose Finding Phase) | Up to 4 years
  The maximum grade of each type of toxicity will be recorded for each patient. For each toxicity reported by dose level, the percentage of patients developing any degree of that toxicity as well as the percentage of patients developing a severe degree (grade 3 or higher) will be determined.

SECONDARY OUTCOMES:
Tolerability (Dose Expansion Phase) | Upon completion of the dose expansion phase
  The maximum grade of each type of adverse event will be recorded for each patient and the percentage of patients developing any degree of that adverse event as well as the percentage of patients developing a severe degree (grade 3 or higher) will be determined.
Tumor response rate (Dose Expansion Phase) | Up to 4 years
  Defined as the number of patients whose tumor has met the immune-modified Response Evaluation Criteria in Solid Tumors criteria for complete response (CR) or partial response (PR) on two consecutive evaluations at least 8 weeks apart among all the eligible patients who have begun treatment. A 90% binomial confidence interval for the tumor response rate will be determined.
Duration of response (Dose Expansion Phase) | From the time measurement criteria are met for CR or PR until the first date that recurrent or progressive disease is objectively documented, assessed up to 4 years
  Will be estimated using the Kaplan-Meier method.
Overall survival (Dose Expansion Phase) | From study entry to death due to any cause, assessed up to 4 years
  Will be estimated using the Kaplan-Meier method.
Progression-free survival (Dose Expansion Phase) | From study entry to the documentation of disease progression, assessed up to 4 years
  Will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto A Leon-Ferre, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (10):
- United States (10):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm